CLINICAL TRIAL: NCT04073849
Title: Evaluation of CD71 Expression in a Dried Blood Spot Following rEPO Administration
Brief Title: CD71 in Dried Blood Spots in Healthy Males
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Sports Medicine Research and Testing Laboratory (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: SMRTL-2018_02
Record Dates: First submitted 2019-07-28; First posted 2019-08-29 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2019-03

CONDITIONS: Healthy Athletes
MeSH Terms: interventions — Epoetin Alfa; Erythropoietin; Saline Solution; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Cohort A to receive active drug Cohort B to receive placebo, (saline)
Who Masked: Participant
Masking Description: Online randomization tool
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort A (Active Comparator): EPOGEN® (epoetin alfa) Study Drug Epoetin Alfa (EPOGEN®) 40 IU / kg dose during boosting phase, delivered s.c.; 8 injections 900 IU dose during microdosing, delivered i.v.; 6 injections
  Interventions: Drug: EPOGEN® (epoetin alfa)
- Cohort B (Sham Comparator): Saline 40 IU / kg dose during boosting phase, delivered s.c.; 8 injections 900 IU dose during microdosing, delivered i.v.; 6 injections
  Interventions: Other: Normal Saline

INTERVENTIONS:
Drug: EPOGEN® (epoetin alfa) — Active drug
  Other Names: erythropoietin, rEPO
  Arms: Cohort A
Other: Normal Saline — Placebo
  Other Names: Saline
  Arms: Cohort B

SUMMARY:
Understand the effect of recombinant EPO (rEPO) boosting and microdosing on the hematological module of the Athlete Biological Passport (ABP)

* Measure the change in CD71 longitudinally in subjects from both cohorts
* Assess whether rEPO administration can be detected in a dried blood spot (DBS) using recent advances in analytical methodologies
* Compare windows of rEPO detection using both Athlete Biological Passport models and direct detection using analytical methods in urine, blood, and DBS

DETAILED DESCRIPTION:
Despite being banned by the World Anti-Doping Agency, blood doping is a common method of performance enhancement used by athletes wishing to gain an unfair advantage over their competition. A common way to achieve this increase is by using erythropoiesis stimulating agents (ESA's), namely recombinant erythropoietin (rEPO). Though laboratory tests have been developed for the direct detection of all known isoforms of exogenously administered ESAs in both urine and blood, athletes have found ways to circumvent these testing measures using techniques such as microdosing.

ELIGIBILITY:
Inclusion Criteria: Active individuals, preferably those that participate regularly in endurance athletics either for sport or for leisure, between the ages of 18 and 45

- Participants should have ferritin > 35 ng/mL and transferrin saturation > 20% at the time of enrollment

Exclusion Criteria: Individuals currently enrolled in a registered testing pool for anti-doping purposes

* Individuals with the intent to compete in sanctioned athletic events during the study period
* Unwillingness to provide urine samples or blood samples
* Not actively exercising
* Individuals who show a high risk for MI/CAD, stroke, CHF, and venous thromboembolism (VTE)., as defined by the Principal Investigator
* Individuals with known drug allergies
* Individuals with EKG abnormalities, as determined by the Principal Investigator
* Individuals who have chronic kidney disease, HIV, cancer, hepatitis B, hepatitis C, or are planning surgery during the study
* Individuals with history of acute or chronic medical or psychiatric condition
* GFR (Creatinine clearance) <60 mL/min
* Ferritin >270 ng/mL
* Individuals who have a baseline hemoglobin concentration greater than 15.5 g/dL or a baseline hematocrit above 47%
* Individuals with blood or iron disorders, including polycythemia, hemochromatosis, anemia, or iron-deficiency anemia
* Individuals with a history of bleeding or bone marrow aplasia
* Individuals who are diabetic or with a history of cardiac or hepatic disease or history of drug abuse

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — male
Enrollment: 24 (Actual)
Dates: Start 2019-07-15 (Actual); Primary Completion 2020-11-15 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
CD71 (transferrin receptor) concentration | 8 months
  CD71 concentration will be measured during and following administration and will be compared to established baseline values from each individual and the study population to understand the changes caused by this dosing pattern of rEPO. These data, especially when comparing to the variability in CD71 in the placebo cohort, may be extrapolated in the anti-doping framework to detect rEPO abuse by athletes.
Hemogloblin concentration | 8 months
  Hemoglobin concentration will be measured during and following administration and will be compared to established baseline values from each individual and the study population to understand the changes caused by this dosing pattern of rEPO
Reticulocyte percentage (Ret%) | 8 months
  Ret% will be measured during and following administration and will be compared to established baseline values from each individual and the study population to understand the changes caused by this dosing pattern of rEPO
Calculated OFF-score | 8 months
  Calculated using the formula: OFF-score = Hgb - 60*√Ret%, OFF-score will be calculated from each collection during and following administration and will be compared to established baseline values from each individual and the study population to understand the changes caused by this dosing pattern of rEPO
Immature reticuocyte fraction | 8 months
  The immature reticulocyte fraction (IRF) will be measured during and following administration and will be compared to established baseline values from each individual and the study population to understand the changes caused by this dosing pattern of rEPO.

SECONDARY OUTCOMES:
Window of detection (detectability time) following rEPO use | 12 months
  The length of time (following both the subcutaneous 'boosting' phase and the intravenous 'microdosing' phase) that rEPO use is evident will be assessed. This will be assessed using different criteria:
  1. Direct detection of the rEPO drug in urine, serum (and/or plasma), and dried blood spots
  2. b. Athlete Biological Passport adaptive model
Analytical detection of rEPO in a dried blood spot | 12 months
  Dried blood spot samples will be extracted and analyzed using analytical techniques (namely SAR-PAGE, SDS-PAGE, IEF-PAGE, or others) employed by the laboratory for the direct detection of rEPO.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Eichner, PhD, Study Director — Sports Medicine Research and Testing Laboratory; Andre Crouch, MD, Principal Investigator — Sports Medicine Research and Testing Laboratory
Locations (1):
- Sports Medicine Research and Testing Laboratory, Salt Lake City, Utah, United States